CLINICAL TRIAL: NCT04579484
Title: Determinants of Acquired Endocrine Resistance in Metastatic Breast Cancer: A Pilot Study
Acronym: ENDO-RESIST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: ENDO-RESIST
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Breast Cancer
Keywords: CDK4/6 inhibitors; endocrine resistance; gut microbiome
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples and fecal samples will be collected at baseline, after 1 month on treatment and on change in treatment due to disease progression. Sampling will coincide with clinic visits.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-center prospective study involving analysis of circulating tumor DNA (ctDNA) and the gut microbiome in patients with metastatic breast cancer on standard of care endocrine therapy with an aromatase inhibitor in combination with an inhibitor of the cyclin-dependent kinases 4 and 6 (CDK 4/6). Up to 20 patients with Estrogen Receptor positive (ER+), Human Epidermal Growth Factor Receptor 2 negative (HER2-) metastatic breast cancer and Eastern Cooperative Oncology Group (ECOG) performance status 0-1 will be enrolled. This study involves the collection and analysis of patient samples and does not involve therapeutic intervention.

DETAILED DESCRIPTION:
Endocrine therapies have been associated with an overall survival benefit in breast cancer and are the preferred initial treatment approach in patients with ER+, HER2- metastatic breast cancer. Unfortunately, resistance to endocrine therapies eventually develops in the metastatic setting and metastatic breast cancer remains an incurable disease. Endocrine resistance may develop as a result of alterations in estrogen signaling and metabolism pathways, which may be modulated by gut bacteria. In addition, genomic profiling of archival tissues and circulating tumor DNA (ctDNA) in ER+ breast cancer has identified multiple somatic molecular alterations that may mediate response to endocrine therapies.

This study is designed to identify markers of endocrine resistance in ctDNA and the gut microbiome in patients with ER+ HER2- metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Sign written and voluntary informed consent
* Histological confirmation of advanced ER positive and HER2 negative breast cancer.
* Adult patients at least 18 years of age
* ECOG performance status equal to 0 or 1
* Able to provide written informed consent
* Must be willing to provide blood for ctDNA analysis on study enrollment and at specified study time points
* Must be willing and able to perform stool sample collection
* Patients must be suitable, as per their treating physician, for initiation of first line endocrine therapy with an aromatase inhibitor and a CDK 4/6 inhibitor for metastatic disease

Exclusion Criteria:

* Prior treatment with CDK 4/6 inhibitors in the neoadjuvant or adjuvant setting
* Use of targeted therapies other than endocrine therapies alone in the neoadjuvant or adjuvant setting
* Relapse on prior endocrine therapy or within 6 months of discontinuation of prior adjuvant endocrine therapy
* History of inflammatory bowel disease, chronic diarrhea or malabsorption syndromes and significant prior bowel resection as judged by the study investigator
* Use of immunosuppressants including steroids within the previous 4 weeks of planned Cycle 1 Day 1 treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with ER positive and HER2 negative metastatic breast cancer planned to initiate on standard of care treatment with an aromatase inhibitor and a CDK 4/6 inhibitor
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-02-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure | 12 months
  Time from first treatment on study (standard of care aromatase inhibitor and a CDK 4/6 inhibitor) until the date of treatment discontinuation

SECONDARY OUTCOMES:
Correlation between specific mutations in ctDNA and in archival tissue samples (where available from prior testing) with time to treatment failure | 12 months
  Identification of mutations in archival tissue samples (where available from prior testing) and sequencing of ctDNA using next generation sequencing panel
Diversity and composition of the gut microbiome in patients with ER+ HER2- metastatic breast cancer | 12 months
  Analysis of the gut microbiome via 16S rRNA sequencing and metagenomic sequencing of fecal samples at baseline and at development of progressive disease
Dietary factors and composition of the gut microbiome | 14 days
  Assessment of food intake via dietary questionnaire and correlation with diversity and composition of the gut microbiome
Overall survival | 2 years
  Time from start of treatment until death

CONTACTS AND LOCATIONS:
Overall Officials: Rossanna C. Pezo, MD/PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No